CLINICAL TRIAL: NCT06396286
Title: Spine Surgery for Lenke 1 Adolescent Idiopathic Scoliosis: a Pilot Study
Brief Title: Spine Surgery for Lenke 1 Adolescent Idiopathic Scoliosis
Acronym: BS23
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BS23
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Scoliosis; Spine Deformity; Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): severe adolescent idiopathic scoliosis Lenke 1
  Interventions: Procedure: single rod

INTERVENTIONS:
Procedure: single rod — surgical correction of severe adolescent idiopathic scoliosis with screws and a single rod.

SUMMARY:
Idiopathic scoliosis of developmental age (AIS) is the most vertebral deformity in the adolescent population, with a prevalence of 1-3%. The treatment of AIS depends on the morphology and extent of the curve and the growth potential residual, can range from simple clinical-radiological monitoring, to the use of braces to, in the most severe cases, correction surgical correction. The indication for surgical correction of AIS depends on the location, extent and flexibility of the scoliotic curve and not least on the patient's age or, better, the skeletal age. The primary goal of surgery is to correcting the deformity by preventing its progression, preserving as many motion segments as possible; secondarily, the surgery aims to restore the coronal and sagittal balance of the spine.

DETAILED DESCRIPTION:
Historically, the first internal fixation system used for the correction and arthrodesis of AIS is the Harrington system. The his implant provided minimal invasion of the canal vertebral canal, providing predictable correction of the deformity vertebral but with limited ability to provide control of the sagittal plane, being unable to effectively derotate the spine. Over the years, implants have been applied "second-generation" vertebrae that allow for fixation spinal by implanting pedicle screws and hooks and are more effective in correcting the curve, achieved through distraction and compression maneuvers (Cotrel-Debousset), up to to direct derotation maneuvers using of uniplanar screws that allow effective reduction of the hump costal. These techniques require the implantation of a higher density of surgical instrumentation, requiring more time surgery, greater intraoperative blood loss, greater greater risk of intraoperative neurological damage, and greater reduction spinal mobility. In addition, in recent years there has been increasing emphasis on emphasizing how lower density of the surgical instrumentation conditions the stiffness and tension of the arthrodesis system, resulting in better postoperative outcomes. Although there is awareness of the importance of reducing the invasiveness of the surgical approach, to date the most frequently adopted for the surgical correction of AIS is the vertebral fusion by instrumented arthrodesis, performed using a posterior approach (posterior spinal fusion - PSF). This technique involves a wide median incision with implantation of screws pedicle screws at the level of the vertebral soma, joined together by means of two longitudinal bars, placed lateral to the line of the spinoses. This surgical technique is invasive and is associated with substantial blood loss, severe postoperative pain, as well as the infectious risk of the surgical site. The choice of vertebral levels to be included in arthrodesis follows the classification according to Lenke, which distinguishes different types of curves. In particular, curves of type Lenke 1 would lend themselves to a less invasive approach because they are structured only at the thoracic level being therefore correctable therefore with a more selective approach. Compared with traditional the single bar has the advantage of treating the spine surgically only halfway, that is, on a single side with respect to the plane of the spinoses, i.e., the cut surgery exposes only the posterior arches of the concavity of the scoliotic curve, this results in less tissue damage, reduces the blood loss and consequently reduces infectious risk and allows early mobilization with reduced post surgery.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosis of AIS;
* Male and female sex;
* Age between 12 and 21;
* Thoracic scoliotic curve, type I according to Lenke's classification;
* Preoperative radiographic range of the main scoliotic curve between 40° and 70° Cobb;
* Reducibility of the curve on bending radiographs by 30%;
* Signature of the informed consent of patients/parents to actively participate in the study and clinical follow-up.

EXCLUSION CRITERIA:

* Scoliosis with an etiology different from AIS;
* pre-operative COBB > 70°;
* Patients already treated surgically for scoliosis;
* Location of the scoliotic curve: Lenke 2-6;
* Patients who do not fall within the parameters described;
* Patients unable to express consent or carry out follow-ups;
* Language barrier;
* Pregnant women.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Spine Correction | at baseline
  The correction of the curvature of the back will be evaluated via x-ray
Spine Correction | at 12 months
  The correction of the curvature of the back will be evaluated via x-ray
Quality of Life 1 | at baseline
  The "Scoliosis Research Society 22" is a multidimensional questionnaire covering the four non-management domains of pain, function, self-image, and mental health (5 items per domain), along with 2 items to assess the patient's satisfaction with management of their deformity
Quality of Life 1 | at 12 months
  The "Scoliosis Research Society 22" is a multidimensional questionnaire covering the four non-management domains of pain, function, self-image, and mental health (5 items per domain), along with 2 items to assess the patient's satisfaction with management of their deformity
Quality of Life 2 | at baseline
  The Oswestry Disability Index (ODI) a patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from back pain.
Quality of Life 2 | at 12 months
  The Oswestry Disability Index (ODI) a patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Result] Lenke LG. Lenke classification system of adolescent idiopathic scoliosis: treatment recommendations. Instr Course Lect. 2005;54:537-42. PMID 15948478
- [Result] Renshaw TS. The role of Harrington instrumentation and posterior spine fusion in the management of adolescent idiopathic scoliosis. Orthop Clin North Am. 1988 Apr;19(2):257-67. PMID 3282199